CLINICAL TRIAL: NCT05114525
Title: Analysis of Patient Understanding of Radiation Therapy Among Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-58571; BRS0122 (Other: OnCore)
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients Who are Anticipated to Receive Definitive Treatment (Experimental)
  Interventions: Behavioral: Survey questionnaire

INTERVENTIONS:
Behavioral: Survey questionnaire — The survey questionnaire will include semi-structured questions about patient demographics and patient understanding of the risks and benefits of radiation, different treatment options, the treatment process, utility of visual aid presentation and information gathering preference using a semi-structured questionnaire

SUMMARY:
The purpose of this study is to conduct a descriptive feasibility study of assessing how patients retain and understand information regarding radiation therapy obtained from an initial consult visit. This study will also pilot the use of visual aids and assess their utility to patients during a consult. The study will provide a baseline to conduct larger studies that will later incorporate additional patient education tools to assess changes in patient understanding of information received in radiation oncology patient consultations.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with non-invasive or invasive breast cancer receiving consultation at the breast radiation oncology clinic for radiotherapy recommendations

Exclusion Criteria:

* Patients under 18 years old or receiving palliative care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
post-consultation telephone questionnaire | 10 days
  assess patient understanding and use of visual aids specifically in radiation oncology consultations

SECONDARY OUTCOMES:
correlations between patient survey score as a measure of patient understanding | 10 days following consultation
  Patients will also be asked to rate the ease of understanding of visual aids provided and their utility in facilitating patient understanding of radiation oncology concepts. It will be analyzed via ANOVA to investigate the association of various factors to the patient's total score. Each participant's interview will be scored based on the following scoring system: Correct"=1point; "Incorrect" = 0 point.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Horst, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No